CLINICAL TRIAL: NCT04250779
Title: Evaluating Efficacy of Smart Device in Assisting With Inhaler Technique and Adherence
Acronym: MOMMIASTHMA1
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Landon Pediatric Foundation (Other)
Collaborators: Cognita Labs LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MOMMIASTHMA1
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-01

CONDITIONS: Asthma; Adherence, Medication; Childhood Asthma
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Research will initially involve collection of data describing the participants' current use of their medication following standard education. Subsequent phases will add audio / haptic coaching to the process of administering medication by MDI, and follow the same participants to determine whether or not there is improvement in technique and adherence to therapy.
  The device will be used with a placebo inhaler (given AFTER the participant's regular medication is taken by standard techniques), to determine how participants use the device, and to identify the most effective coaching interventions for this age group. This is to ensure that the device does not interfere with delivery of routine asthma controller medications. The data will be used to develop a subsequent, longer term study in which we will evaluate the effect of the coaching device on asthma control, when it is used with the subject's controller medication.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): In this arm, patients are provided with standard-of-care instructions on using MDIs correctly and regularly at home. The MDI usage is recorded using CapMedic device with active guidance turned off.
  Interventions: Behavioral: Video-based guidance
- Treatment Group (Active Comparator): In this arm, patients are provided with active guidance from CapMedic device on using MDIs correctly and regularly at home. The MDI usage is recorded using CapMedic device with active guidance turned on.
  Interventions: Device: CapMedic smart inhaler device

INTERVENTIONS:
Device: CapMedic smart inhaler device — The CapMedic device provides active coaching to promote correct and regular use of MDI.
  Arms: Treatment Group
Behavioral: Video-based guidance — Patients are shown a video of how to use inhalers correctly and any questions are answered by the clinician. They are also encouraged to use inhalers regularly and correctly at home.
  Arms: Control Group

SUMMARY:
Asthma affects over 10 million children in the U.S., and poses a significant health and cost burden. Metered dose inhaler (MDI) is the most common method of treatment. Studies show that up to 80% of patients demonstrate incorrect use of MDIs, which results in suboptimal medication delivery to the lungs.

Asthma control can be followed by symptoms, rescue medication usage and measures of airflow obstruction. Current options to monitor control include an asthma diary (relies on consistent use by the patient), pharmacy records of medication dispensing (dispensing does not equal usage), and peak expiratory flow (PEF) meters (significant variability in technique leading to inconsistent results).

CapMedic is a smart inhaler and home spirometer device which aims to assist with correct MDI usage and to monitor asthma control. CapMedic fits on top of the MDI inhaler and provides live audio-visual-haptic cues to guide the patient for correctly using their inhaler. CapMedic includes a built-in forced expiratory flow in 1 second (FEV1, a measure of airflow) and PEF meter. It will utilize the same audio-visual-haptic hardware to implement live cues that encourage patient's effort in performing accurate at-home FEV1/PEF test. Cap will also be able to log medication usage and Medic application will allow patients to keep an asthma symptom diary.

DETAILED DESCRIPTION:
CapMedic is a smart inhaler and home spirometer device which aims to assist with correct MDI usage and to monitor asthma control. CapMedic fits on top of the MDI inhaler and provides live audio-visual-haptic cues to guide the patient for correctly using their inhaler. CapMedic includes a built-in forced expiratory flow in 1 second (FEV1, a measure of airflow) and PEF meter. It will utilize the same audio-visual-haptic hardware to implement live cues that encourage patient's effort in performing accurate at-home FEV1/PEF test. Cap will also be able to log medication usage and Medic application will allow patients to keep an asthma symptom diary.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Asthma
* Regular user of MDI
* Asthma Control Test (ACT) scores between 15 and 25
* FEV1 between 60-80% of predicted (persistent mild-moderate)
* Disease severity in the range mild-moderate
* Access to a Smartphone and internet during the entire duration of the study.
* Cognitively able to utilize the device and express interest in participating.

Exclusion Criteria:

* Patients without asthma
* With developmental disabilities
* Do not speak English
* Do not own a Smartphone

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
MDI use Competence in Clinic | 1 day
  Correctness of Inhaler Use measured using CapMedic device during recruitment. Competence is measured as a score out of 4 for 4 steps of MDI use: 1. Shaking, 2. Orientation, 3. Coordination 4. Duration of inhalation
MDI use Competence at home | 8 weeks
  Correctness of Inhaler Use measured using CapMedic device at home. Competence is measured as a score out of 4 for 4 steps of MDI use: 1. Shaking, 2. Orientation, 3. Coordination 4. Duration of inhalation

SECONDARY OUTCOMES:
PEF Lung Function in Clinic | 1 day
  PEF measured using CapMedic device during recruitment. PEF is measured in L/min.
FEV1 Lung Function in Clinic | 1 day
  FEV1 measured using CapMedic device during recruitment. FEV1 is measured in L.
PEF Lung Function at home | 8 weeks
  PEF measured using CapMedic device at home. PEF is measured in L/min.
FEV1 Lung Function at home | 8 weeks
  FEV1 measured using CapMedic device at home. FEV1 is measured in L.
MDI use Adherence | 8 weeks
  Regularity of MDI use measured by CapMedic device at home, measured as a % of puffs taken per week compared to prescribed dosage.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Diagnostic Center, Ventura, California, United States

REFERENCES:
- [Derived] Chan A, De Simoni A, Wileman V, Holliday L, Newby CJ, Chisari C, Ali S, Zhu N, Padakanti P, Pinprachanan V, Ting V, Griffiths CJ. Digital interventions to improve adherence to maintenance medication in asthma. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD013030. doi: 10.1002/14651858.CD013030.pub2. PMID 35691614